CLINICAL TRIAL: NCT03007459
Title: The Health of Competitive Fitness Athletes, a Cohort Study of Female Fitness Athletes and Physical Active Control's During and After Three Months of Fitness Contest Dieting
Brief Title: The Health of Competitive Fitness Athletes
Status: Completed | Type: Observational
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: 3281
Record Dates: First submitted 2016-12-24; First posted 2017-01-02 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Resting Metabolic Rate; Bone Mineral Density, Low, Susceptibility to; Body Image; Perfectionism; Depression; Eating Disorder; Exercise-Related Amenorrhea; Exercise Addiction; Binge Eating; Dietary Amenorrhea; Dietary Deficiency
Keywords: Body composition; Bone mineral density; Binge Eating; Eating Disorder; Exercise Dependency; Depression; Perfectionism; Body building; Drive for Muscularity; Drive for leanness
MeSH Terms: conditions — Depression; Feeding and Eating Disorders; Bulimia; Malnutrition | interventions — Mental Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Female Fitness Athletes: Psychological health and physiological health of fitness athletes
  Interventions: Other: Psychological health; Other: Physiological health
- Female, physically active Controls: Psychological health and physiological health of female controls
  Interventions: Other: Psychological health; Other: Physiological health

INTERVENTIONS:
Other: Psychological health — Observing and measuring baseline, and changes in, psychological health through a fitness contest preparation period
Other: Physiological health — Observing and measuring baseline, and changes in, physiological health through a fitness contest preparation period

SUMMARY:
Fitness athletes emphasize the value of staying lean, muscular and defined, and motivates and inspires followers through social media. We want to study the effect of such lifestyle on selected aspects of psychological and physical health in female fitness athletes, and compare the outcomes to a healthy, physically active female population.

DETAILED DESCRIPTION:
Little is known about the mental and physical health effect from following the modern, idealized fitness lifestyle. The lifestyle is characterized by selective and restrictive eating behavior, strength training and use of supplements. The athletes emphasize the value of staying lean, muscular and defined, and motivates and inspires followers through social media. This study will recruit and observe a group of competitive female fitness athletes over their typical 3 month dieting period when preparing for contest. Before their contest diet is initiated, the athletes will be screened on selected aspects of psychological and physical health. The screening is repeated two weeks prior to their first seasonal contest, and then finally one month post-contest season. During the diet period of 3 months, the athletes answers brief questionnaires by email on eating- and training behavior and on mood, while also reporting dietary intake by telephone interview.

Recreational physically females, not planning to do any fitness contest, will be recruited to serve as a parallel control group. They will perform the same physical and psychological screening, and answer the same questionnaires throughout the fitness contest diet period.

ELIGIBILITY:
Inclusion Criteria:

* Fitness athletes: planning to compete in fitness sport during spring or fall 2017
* Controls: being regular physically active (exercise >2 times/week during last year) with a BMI between 17,5-30

Exclusion Criteria:

* Controls: having competed in fitness sports previously or planning to do in the future, or working as a personal trainer.
* Not able to meet at the Norwegian School of Sport Sciences for baseline and follow up screenings.
* Being pregnant or nursing
* Metabolic related diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female, fitness athletes are being recruited through social media, Fitness team leaders and the Norwegian national federation for Bodybuilding and Fitness.
  Physically active, female controls are being recruited through social media, training facilities and through colleagues at the Norwegian School of Sport Sciences
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Body composition | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to post-test, for lean body mass and fat mass, measured with Dual Xray absorptiometry (DXA)

SECONDARY OUTCOMES:
Resting Metabolic Rate | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to posttest, for resting metabolic rate, measured with indirect calorimetry
Bone Mineral Density | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to post-test, for bone mineral density measured with Dual Xray absorptiometry (DXA)
Perfectionism | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Comparing scores on perfectionism between case and controls, and individual changes in scores through study period, with Child Adolescent Perfectionism Scale (CAPS 22 items)
Depression | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to post-test, for scores on depressive mood, measured with Becks Depression Inventory (BDI)
Eating disorders | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to post-test, for scores on Eating disorder examination questionnaire (EDE-q)
Eating behavior; binge eating | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to post-test, for scores on Binge Eating Scale (BES)
Eating behavior; restrictive eating and sensation of hunger | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline values, change from pre-test to mid-test, and finally change from mid- to post-test, for scores on Three Factor Eating Questionnaire (TFEQ-21)
Menstrual Status, self-reported | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline status, change from pre-test to mid-test, and finally change from mid- to post-test, for self-reported menstruation health (Low Energy Availability in Females questionnaire, LEAF)
Dietary intake, weighed diet registration | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Change in dietary intake. Baseline status, change from pre-test to mid-test, and finally change from pre- to post-test, evaluated with weighed dietary registration and analysed with national analytical software (Kostholdsplanleggeren.no)
Exercise dependency | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline status, change from pre-test to mid-test, and finally change from pre- to post-test, evaluated with Exercise Dependency Scale (EDS)
Reason for Exercise | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline status, change from pre-test to mid-test, and finally change from pre- to post-test, evaluated with Reason for Exercise Inventory (REI)
Depression | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Changes in reported state of depression during the dieting period of fitness athletes, measured with BDI
Dietary intake, 24-hour recall interview | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Changes in energy and nutrient intake during the dieting period of fitness athletes, measured with dietary 24-hour recall interview and analysed with national analytical software (Kostholdsplanleggeren.no)
Menstrual cycle, self reported | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Self reported menstrual bleeding's during the dieting period of fitness athletes (LEAF)
Eating disordered behavior | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Changes in eating behavior during the dieting period of fitness athletes, measured with the behavioral aspects of EDE-q
Eating behavior; binge eating behavior | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Changes in eating behavior during the dieting period of fitness athletes, measured with BES
Eating behavior; restrictive eating and sensation of hunger | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Changes in eating behavior during the dieting period of fitness athletes, measured with TFEQ-21
Training volume, self reported | Each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Reporting number of training sessions pr week and type of exercise (endurance related exercise or strength training)
Training history, self reported | Retrospective
  Reporting experience with training, giving details on specific sport activity and typical intensity
Dietary Supplements | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest), and each 2nd week during the 3 month contest dieting period (between pre-test and mid-test)
  Reporting usage of dietary supplements during the dieting period
Eating disorders, history | Retrospective
  Reporting previous eating disorder and whether treatment were recieved or not
Drive for Muscularity | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline status, change from pre-test to mid-test, and finally change from pre- to post-test, evaluated with Drive for Muscularity (DM) (McCreary & Sasse 2000)
Drive for Leanness | Pre-test (3 months before contest), mid-test (2 weeks before contest) and post-test (one month post-contest)
  Baseline status, change from pre-test to mid-test, and finally change from pre- to post-test, evaluated with Drive for Leanness (DL) (Smolak & Murnen 2008)
Body Weight, history | Retrospective
  Reporting lowest and highest bodyweight after 18 yr's of age (excluding periods of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn K Sundgot-Borgen, Professor, Study Director — Professor
Locations (1):
- Norwegian School of Sports Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not planned to be available to other than the research group.

REFERENCES:
- [Derived] Mathisen TF, Engen KM, Sundgot-Borgen J, Stensrud T. Evaluation of a short protocol for indirect calorimetry in females with eating disorders and healthy controls. Clin Nutr ESPEN. 2017 Dec;22:28-35. doi: 10.1016/j.clnesp.2017.09.003. Epub 2017 Oct 5. PMID 29415831